CLINICAL TRIAL: NCT02946073
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Enriched-Enrollment Withdrawal, Multicenter Study to Evaluate the Efficacy and Safety of a Long-Acting Subcutaneous Injectable Depot of Buprenorphine (CAM2038) in Subjects With Moderate to Severe Chronic Low Back Pain Currently Treated With Daily Opioids
Brief Title: Buprenorphine (CAM2038) in Subjects With a Recent History of Moderate to Severe Chronic Low Back Pain
Acronym: CAM2038
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braeburn Pharmaceuticals (Industry)
Collaborators: Medpace, Inc. (Industry); Camurus AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-16-555
Record Dates: First submitted 2016-10-07; First posted 2016-10-26 (Estimated); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-01

CONDITIONS: Chronic Lower Back Pain; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): CAM2038 placebo injections
  Interventions: Other: Placebo
- CAM2038 (Experimental): CAM2038 50 mg/mL q1w at doses of 8 mg, 12 mg, 16 mg, 24 mg, or 32 mg. CAM2038 356 mg/mL q4w at doses of 64 mg, 96 mg, or 128 mg.
  Interventions: Drug: buprenorphine

INTERVENTIONS:
Drug: buprenorphine
  Other Names: CAM2038
  Arms: CAM2038
Other: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase III, placebo-controlled, multicenter study with an enriched-enrollment withdrawal (EEW) design to evaluate the efficacy and safety of CAM2038 in opioid-experienced subjects with moderate to severe CLBP that requires continuous, around-the-clock (ATC) opioid treatment ≥ 40 mg morphine equivalent dose (MED). The study includes 5 phases: A Screening Phase (up to 2 weeks), a Transition Phase (up to 2 weeks), an Open-Label Titration Phase (up to 10 weeks), a Double-Blind Treatment Phase including a Final Study Visit (12 weeks), and a Follow-up Phase (4 weeks). The overall duration of participation in the core phase of the study (randomized Double-Blind Phase) is up to 30 weeks, from the Screening Phase through the Follow-up Phase. Subjects who complete the Double-Blind Treatment Study Phase will be offered an opportunity to continue treatment in an open label safety extension for up to 60 weeks. Additional subjects may be recruited to open label safety extension to meet the goal of 100 subjects with 60 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided prior to the conduct of any study-related procedures.
2. Male or non-pregnant, non-lactating female subject, greater than or equal to 18 years old.
3. Body mass index (BMI) between 18 and 38 kg/m2, inclusive.
4. Treated with daily opioids for moderate to severe CLBP for a minimum of 3 months prior to Screening.
5. On a stable dose of ≥40 mg/day of oral morphine or MED during the 14 days prior to Screening.
6. Systolic blood pressure ≥100 mmHg and diastolic blood pressure ≥60 mmHg.
7. Female subject of childbearing potential who is willing to use a reliable method of contraception during the entire study (Screening Visit to final Follow-up). To be considered not of childbearing potential, female subjects must be surgically sterile (hysterectomy or bilateral oophorectomy, or bilateral tubal ligation with surgery at least 6 weeks before Screening).
8. Male subject who is willing to use reliable contraception
9. Willing and able to comply with all study procedures and requirements.

Exclusion Criteria:

1. Positive for hepatitis B surface antigen, hepatitis C viral RNA, or antibodies to human immunodeficiency virus (HIV).
2. Clinically significant symptoms, medical conditions, or other circumstances which, in the opinion of the investigator, would preclude compliance with the protocol, adequate cooperation in the study, or obtaining informed consent, or may prevent the subject from safely participating in the study, including the following:

   1. Severe respiratory insufficiency, respiratory depression, airway obstruction, gastrointestinal motility disorders, biliary tract disease, severe hepatic insufficiency, or planned surgery.
   2. Bipolar disorder
3. Current diagnosis of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition-defined moderate to severe substance use disorder (including alcohol), other than caffeine or nicotine.
4. Female subject planning to become pregnant during the study.
5. Surgical procedure(s) for CLBP within 6 months prior to Screening.
6. Concomitant disease(s) that could prolong the QTcF interval, such as autonomic neuropathy (caused by diabetes or Parkinson's disease), HIV, cirrhosis, Long QT Syndrome, or family history of Long QT Syndrome.
7. QTcF >450 ms for males and >470 ms for females, or clinically significant electrocardiogram (ECG) abnormality at Screening, at the investigator's discretion.
8. Currently taking medications that have the potential to prolong the QTcF interval or may require such medications during the course of the study (Appendix 1) and has clinically significant abnormalities on screening ECG readings, as determined by the investigator.
9. A nerve or plexus block, including epidural steroid injections or facet blocks, within 1 month prior to Screening or botulinum toxin injection in the lower back region within 3 months of Screening.
10. History of chemotherapy or confirmed malignancy (except basal cell carcinoma) within the past 2 years.
11. Any other acute or chronic pain condition that could interfere with the subject's ability to report their CLBP accurately and consistently and/or interfere with the study staff's ability to assess the subjects CLBP.
12. An active or pending workman's compensation, insurance claim, or litigation related to back pain (i.e., primary claim is back pain).
13. Clinically significant history, in the opinion of the investigator, of suicidal ideation or current evidence that the subject is actively suicidal.
14. Clinically significant history of major depressive disorder that is poorly controlled with medication, per investigator judgment.
15. Hypersensitivity or allergy to BPN, other opioids, or excipients of CAM2038.
16. Hypersensitivity or allergy to acetaminophen.
17. Use of strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4), such as some azole antifungals (e.g., ketoconazole), macrolide antibiotics (e.g., clarithromycin), or protease inhibitors (e.g., ritonavir, indinavir, and saquinavir) within the 30 days prior to Screening,
18. Use or planned use of natural supplements that can affect CYP3A4, such as St. John's Wort, throughout the study.
19. Has a major bleeding disorder, such as hemophilia, or treated with high levels of anticoagulants per the investigator's discretion.
20. Current or confirmed past diagnosis of Sphincter of Oddi dysfunction.
21. Has a significant hepatic disease, as indicated by Screening clinical laboratory assessment results (aspartate aminotransferase, alanine aminotransferase, or lactate dehydrogenase values ≥3 × the upper limit of normal [ULN]) or has a creatinine value ≥1.5 × ULN).
22. Is an employee of the investigator or the trial site, with direct involvement in the proposed trial or other studies under the direction of the investigator or trial site or is a family member of the investigator or of an employee of the investigator.
23. Has any pending legal action that could prohibit participation or compliance in the study.

Criteria for Entry into the Titration Phase:

1. After at least a 12-hour washout from the last IR morphine dose, subject must have a COWS ≥5 and an API pain score over the past 24 hours ≥5 in order to receive a test dose of Buprenex.
2. Passed all baseline criteria, including a normal QTcF, had no change in QTcF >30 ms at 1 hour after the test dose with Buprenex, and had a COWS score <5 after the test dose with Buprenex.

Note:

* Subjects on BPN at Screening are required to participate in the down titration and will undergo a washout period prior to the test dose and first on-study treatment. Subjects entering the study on BPN will not transition to IR Morphine, but will refrain from taking their BPN for 12 -24 hours prior to the test dose to achieve the desired washout period.
* Subjects on BPN at Screening are still required to follow the same Day 1 procedures (e.g., confirmation of pain scores, COWS assessment and Buprenex test dose) as non-BPN subjects.

Criteria for Randomization into the Double-Blind Phase:

1. Been on a stable dose of CAM2038 q1w for at least 2 consecutive weeks.
2. CAM2038 titrated to a dose that provides analgesia (i.e., 7-day API score of ≤4 and at least 2 points below the value at the start of Titration Phase) and is well tolerated for 7 days before randomization.
3. Requires no more than an average of one hydrocodone/acetaminophen 5 mg/325 mg/day during the last 7 days prior to randomization.
4. Demonstrated study medication (CAM2038) compliance ≥80% during the previous 14 days.
5. Demonstrated daily compliance with pain intensity scoring for ≥11 of the previous 14 days, including the last 3 days prior to randomization.

Inclusion Criteria for Open Label Extension For Subjects Continuing from The Randomized Double-Blind Phase.

Subjects must have:

1. Completed Double Blind Phase of the study
2. Signed Informed Consent for Safety Extension

Subjects completing the double-blind phase will be enrolled directly into the open label extension at their respective dose level of CAM2038. They will not be required to participate in a Buprenex treatment test dosing or participate in a titration phase.

For De Novo Subjects (New Subjects Recruited Directly into The Open Label Extension)

Subjects who are not participating in the Double-Blind Phase of the Study must meet all of the following inclusion criteria in order to be eligible for participation in the study:

1. Written informed consent provided prior to the conduct of any study-related procedures.
2. Male or non-pregnant and non-lactating female subject, greater than or equal to 18 years old.
3. BMI between 18 and 38 kg/m2, inclusive.
4. Treated with daily opioids for moderate to severe chronic pain disorder such as CLBP or osteoarthritis for a minimum of 3 months prior to Screening.
5. On a stable dose of >40 mg/day of oral morphine or MED during the 14 days prior to Screening.
6. Systolic blood pressure ≥100 mmHg and diastolic blood pressure ≥60 mmHg.
7. Female subject of childbearing potential who is willing to use a reliable method of contraception during the entire study (Screening Visit to final Follow-up). To be considered not of childbearing potential, female subjects must be surgically sterile (hysterectomy or bilateral oophorectomy, or bilateral tubal ligation with surgery at least 6 weeks before Screening).
8. Male subject who is willing to use reliable contraception
9. Willing and able to comply with all study procedures and requirements.

Exclusion Criteria for Subjects Continuing from The Randomized Double-Blind Phase

1. Clinically significant symptoms, medical conditions, or other circumstances which, in the opinion of the investigator, would preclude compliance with the protocol, adequate cooperation in the study, or obtaining informed consent, or may prevent the subject from safely participating in the study.

Exclusion Criteria for De Novo Subjects only:

Same exclusion criteria as for subjects participating in the Randomized Double-Blind Treatment Phase.

Criteria for Entry into the Titration Phase (for De novo subjects):

1. After at least a 12-hour washout from the last IR morphine dose, subject should have a COWS ≥5 and an API pain score over the past 24 hours ≥5 in order to receive a test dose of Buprenex.
2. Passed all baseline criteria, including a normal QTcF, had no change in QTcF >30 ms at 1 hour after the test dose with Buprenex, and had a COWS score <5 after the test dose with Buprenex.

Note:

* Subjects on BPN at Screening are required to participate in the down titration and will undergo a washout period prior to the test dose and first on-study treatment. Subjects entering the study on BPN will not transition to IR Morphine, but will refrain from taking their BPN for 12 -24 hours prior to the test dose to achieve the desired washout period.
* However, subjects on BPN at Screening are still required to follow the same Day 1 procedures (e.g., confirmation of pain scores, COWS assessment and Buprenex test dose) as non-BPN subjects.

Criteria for Enrolment into the Open Label Treatment Phase (for de Novo subjects):

1. Been on a stable dose of CAM2038 q1w for at least 2 consecutive weeks.
2. CAM2038 titrated to a dose that provides analgesia (i.e., 7-day API score of ≤4 and at least 2 points below the value at the start of Titration Phase) and is well tolerated for 7 days before randomization.
3. Requires no more than an average of one hydrocodone/acetaminophen 5 mg/325 mg/day during the last 7 days prior to randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- United States (69):
  - Parkway Medical Center, Birmingham, Alabama
  - Boyett Health Services Inc, Hamilton, Alabama
  - National Centers for Pain Management and Research, Vestavia Hills, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Phoenix Clinical, Phoenix, Arizona
  - Noesis Pharma, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - MD Studies, Inc., Fountain Valley, California
  - Neuro-Pain Medical Center, Fresno, California
  - Alliance Research Centers, Laguna Hills, California
  - Clinical Trials Research, Lincoln, California
  - Catalina Research Institute, LLC, Montclair, California
  - Allied Clinical Research, LLC, Sacramento, California
  - Care Practice, San Francisco, California
  - Syrentis Clinical Research, Santa Ana, California
  - Universal Pain Management Group, Valencia, California
  - Tampa Pain Relief Center-Brandon, Brandon, Florida
  - International Research Partners, Doral, Florida
  - Dr. Vijapura and Associates, Jacksonville, Florida
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Lake Howell Health Center, Maitland, Florida
  - Ocean Blue Medical Research Center, Inc., Miami Springs, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - FMPM Research, St. Petersburg, Florida
  - Clinical Research of West Florida-Tampa, Tampa, Florida
  - Tampa Pain Relief Centers-Hillsborough, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - River Birch Research Alliance LLC, Blue Ridge, Georgia
  - Columbus Regional Research Institute, Knoxville, Georgia
  - Drug Studies America, Marietta, Georgia
  - Non-Surgical Orthopedics, P.C., Marietta, Georgia
  - Injury Care Research, LLC, Boise, Idaho
  - Millennium Pain Center, Bloomington, Illinois
  - Clinical Investigation Specialists, Inc.-Gurnee, Gurnee, Illinois
  - Medisphere Medical Research Center, Evansville, Indiana
  - International Clinical Research Institute Inc., Overland Park, Kansas
  - Phoenix Medical Research, Prairie Village, Kansas
  - Otrimed, Edgewood, Kentucky
  - River Cities Clinical Research Center, Shreveport, Louisiana
  - Boston Paincare, Waltham, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Amicis Trials, Festus, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - New York Clinical Trials, Inc, New York, New York
  - MedEx Healthcare Research, Inc-NY, New York, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Rapha Institute for Clinical Research, Fayetteville, North Carolina
  - OnSite Clinical Solutions, LLC-Hickory, Hickory, North Carolina
  - Center for Clinical Research, LLC-Winston-Salem, Winston-Salem, North Carolina
  - Aventiv Research, Inc., Columbus, Ohio
  - Dayton Outpatient Center (DOC) Clinical Research, Dayton, Ohio
  - Providence Health Partners-Center for Clinical Research, Dayton, Ohio
  - Medical Research Internationl, Oklahoma City, Oklahoma
  - SP Research, PLLC, Oklahoma City, Oklahoma
  - Frost Medical Group, LLC, Conshohocken, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Coastal Carolina Research Center, Charleston, South Carolina
  - Medical Research South, LLC, Charleston, South Carolina
  - New Phase Research & Development, Knoxville, Tennessee
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Renaissance Clinical Research and Hypertension Clinic, Dallas, Texas
  - Research Concepts GP, LLC-Houstion, Houston, Texas
  - Pioneer Research Solutions Inc., Houston, Texas
  - The Pain Relief Center, Plano, Texas
  - The SMART Clinic/Physicians Research Options LLC, Draper, Utah
  - EPIC Medical Research, Murray, Utah
  - Aspen Clinical Research, Orem, Utah
  - Mid Columbia Research, Richland, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 965 of those subjects entered the Double Blind phase of the study. 108 subjects signed consent as De Novo subjects, but 20 of those subjects were part of the Double Blind phase. The total number of subjects that signed consent was 1053 (965 + 88).Two sites had quality issues with the data, so those subjects were eliminated from the analysis. This made the total number of subjects who were analyzed 222 in the double blind randomized phase and 132 subjects for the open label phase.
Pre-assignment Details: Subjects are screened prior to entry into a titration phase where they are titrated to an appropriate dose. Once they are titrated, they were randomized and entered the double blind period or open label period for de novo subjects.
Groups:
- CAM2038 q1w or q4w BPN Treatment- Double Blind Phase: CAM2038 50 mg/mL q1w at doses of 8 mg, 12 mg, 16 mg, 24 mg, or 32 mg. CAM2038 356 mg/mL q4w at doses of 64 mg, 96 mg, or 128 mg. buprenorphine
- Placebo Subcutaneous Injections-Double Blind Phase: CAM2038 placebo: 0.16, 0.18, 0.24, 0.27, 0.36, and 0.64 mL SC injection administered once weekly or once monthly
- De Novo Subjects-Open Label Phase: De Novo subjects proceeded directly from the Open-Label Titration Period to the Open-Label Safety Extension Phase without participating in the Double-Blind Treatment Period. CAM2038 q1w (buprenorphine FluidCrystal®) : SC injection depot for once weekly or monthly administration at doses of 4, 8, 12, 16, 24 and 32 mg (buprenorphine base) 0.16, 0.24, and 0.64 mL SC injection CAM2038 (buprenorphine FluidCrystal® once-weekly injection depot)
  CAM2038 q4w ( buprenorphine FluidCrystal®): SC injection depot for once monthly administration (356 mg/mL) at doses of 64, 96, 128 or 160 mg (buprenorphine base) 0.18, 0.27, and 0.36 mL SC injection CAM2038 (buprenorphine FluidCrystal® once-monthly injection depot)
- Rollover Subjects-Open Label: CAM2038 q1w (buprenorphine FluidCrystal®) : SC injection depot for once weekly or monthly administration at doses of 4, 8, 12, 16, 24 and 32 mg (buprenorphine base) 0.16, 0.24, and 0.64 mL SC injection CAM2038 (buprenorphine FluidCrystal® once-weekly injection depot)
  CAM2038 q4w ( buprenorphine FluidCrystal®): SC injection depot for once monthly administration (356 mg/mL) at doses of 64, 96, 128 or 160 mg (buprenorphine base) 0.18, 0.27, and 0.36 mL SC injection CAM2038 (buprenorphine FluidCrystal® once-monthly injection depot)
Period: Titration Phase
Arm/Group | CAM2038 q1w or q4w BPN Treatment- Double Blind Phase | Placebo Subcutaneous Injections-Double Blind Phase | De Novo Subjects-Open Label Phase | Rollover Subjects-Open Label
Started (Subjects were not randomized at this time, so all were receiving open-label CAM2038.) | 811 | 0 | 98 | 0
Completed (Subjects were not randomized at this time, so all were receiving open-label CAM2038.) | 222 | 0 | 75 | 0
Not Completed | 589 | 0 | 23 | 0
Period: Double Blind Phase
Arm/Group | CAM2038 q1w or q4w BPN Treatment- Double Blind Phase | Placebo Subcutaneous Injections-Double Blind Phase | De Novo Subjects-Open Label Phase | Rollover Subjects-Open Label
Started | 112 | 110 | 0 | 0
Completed | 88 | 70 | 0 | 0
Not Completed | 24 | 40 | 0 | 0
Period: Open Label Phase
Arm/Group | CAM2038 q1w or q4w BPN Treatment- Double Blind Phase | Placebo Subcutaneous Injections-Double Blind Phase | De Novo Subjects-Open Label Phase | Rollover Subjects-Open Label
Started | 0 | 0 | 75 | 57
Completed | 0 | 0 | 54 | 44
Not Completed | 0 | 0 | 21 | 13

BASELINE CHARACTERISTICS:
Groups:
- Placebo Subcutaneous Injections-Double Blind Phase: CAM2038 placebo: 0.16, 0.18, 0.24, 0.27, 0.36, and 0.64 mL SC injection administered once weekly or once monthly (matching volumes for CAM2038 q1w and near-matching volumes for CAM2038 q4w).
- De Novo Subjects-Open Label; Rollover Subjects-Open Label: CAM2038 q1w (buprenorphine FluidCrystal®) : SC injection depot for once weekly or monthly administration at doses of 4, 8, 12, 16, 24 and 32 mg (buprenorphine base) 0.16, 0.24, and 0.64 mL SC injection CAM2038 (buprenorphine FluidCrystal® once-weekly injection depot)
  CAM2038 q4w ( buprenorphine FluidCrystal®): SC injection depot for once monthly administration (356 mg/mL) at doses of 64, 96, 128 or 160 mg (buprenorphine base) 0.18, 0.27, and 0.36 mL SC injection CAM2038 (buprenorphine FluidCrystal® once-monthly injection depot)
- Total: Total of all reporting groups
Arm/Group | CAM2038 q1w or q4w BPN Treatment- Double Blind Phase | Placebo Subcutaneous Injections-Double Blind Phase | De Novo Subjects-Open Label | Rollover Subjects-Open Label | Total
Number analyzed (Participants) | 112 | 110 | 75 | 57 | 354
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Double Blind Phase Only
  years
    number analyzed (Participants) | 112 | 110 | 0 | 0 | 222
    (all) | 53.7 (12.19) | 54.7 (11.36) |  |  | 54.2 (11.77)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Open Label Phase Only
  years
    number analyzed (Participants) | 0 | 0 | 75 | 57 | 132
    (all) |  |  | 54.3 (10.27) | 56.4 (11.49) | 55.2 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Double Blind Phase only.
  Participants
    number analyzed (Participants) | 112 | 110 | 0 | 0 | 222
    Female | 66 | 56 |  |  | 122
    Male | 46 | 54 |  |  | 100
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Open Label Phase Only
  Participants
    number analyzed (Participants) | 0 | 0 | 75 | 57 | 132
    Female |  |  | 44 | 34 | 78
    Male |  |  | 31 | 23 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Double Blind Phase Only
  Participants
    number analyzed (Participants) | 112 | 110 | 0 | 0 | 222
    Hispanic or Latino | 11 | 11 |  |  | 22
    Not Hispanic or Latino | 101 | 97 |  |  | 198
    Unknown or Not Reported | 0 | 2 |  |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Open Phase Only
  Participants
    number analyzed (Participants) | 0 | 0 | 75 | 57 | 132
    Hispanic or Latino |  |  | 1 | 4 | 5
    Not Hispanic or Latino |  |  | 73 | 51 | 124
    Unknown or Not Reported |  |  | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Double Blind Phase Only
  Participants
    number analyzed (Participants) | 112 | 110 | 0 | 0 | 222
    American Indian or Alaska Native | 1 | 0 |  |  | 1
    Asian | 0 | 1 |  |  | 1
    Native Hawaiian or Other Pacific Islander | 1 | 0 |  |  | 1
    Black or African American | 10 | 12 |  |  | 22
    White | 100 | 97 |  |  | 197
    More than one race | 0 | 0 |  |  | 0
    Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Open Label Phase Only
  Participants
    number analyzed (Participants) | 0 | 0 | 75 | 57 | 132
    American Indian or Alaska Native |  |  | 1 | 0 | 1
    Asian |  |  | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander |  |  | 1 | 0 | 1
    Black or African American |  |  | 6 | 7 | 13
    White |  |  | 67 | 49 | 116
    More than one race |  |  | 0 | 0 | 0
    Unknown or Not Reported |  |  | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. Population: Double Blind Phase Only
  kg/m^2
    number analyzed (Participants) | 112 | 110 | 0 | 0 | 222
    (all) | 29.1 (4.78) | 29.3 (5.27) |  |  | 29.2 (5.02)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. Population: Open Label Phase Only
  kg/m^2
    number analyzed (Participants) | 0 | 0 | 75 | 57 | 132
    (all) |  |  | 29.5 (5.55) | 29.1 (5.29) | 29.3 (5.42)
Pain Score at Start of Open-Label Titration Period [Mean (Standard Deviation); unit: units on a scale] — 11- Point Numerical Rating Scale (NRS-11)- an 11-point scale with anchors at 0 (no pain) and 10 (worst pain imaginable) to measure pain. Population: Double Blind Phase Only
  units on a scale
    number analyzed (Participants) | 112 | 110 | 0 | 0 | 222
    (all) | 7.0 (1.42) | 7.0 (1.39) |  |  | 7.0 (1.40)
Pain Score at Start of Open-Label Titration Period [Mean (Standard Deviation); unit: units on a scale] — 11- Point Numerical Rating Scale (NRS-11)- an 11-point scale with anchors at 0 (no pain) and 10 (worst pain imaginable) to measure pain. Population: Open Label Phase Only
  units on a scale
    number analyzed (Participants) | 0 | 0 | 75 | 57 | 132
    (all) |  |  | 6.7 (1.46) | 6.6 (1.73) | 6.7 (1.57)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Average of (Daily) Average Pain Intensity (WAAPI) and the Primary Timepoint Will be Week 12 of the Double-Blind Phase.
Description: Change from baseline in Weekly Average of (Daily) Average Pain Intensity (WAAPI) and the primary timepoint will be Week 12 of the Double-Blind Phase based on the 11-Point numerical rating scale with 0 being no pain and 10 being the worst pain.
Time Frame: 12 weeks- from randomization baseline to 12 weeks after randomization
Population: Modified Intent-to-Treat (mITT) Population: The mITT Population consisted of all randomized subjects, with the exception of the subjects from Sites 068 and 077 due to persistent site non-compliance
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CAM2038 (Buprenorphine FluidCrystal®) q1w and q4w: CAM2038 q1w (buprenorphine FluidCrystal®) : SC injection depot for once weekly or monthly administration at doses of 4, 8, 12 mg (buprenorphine base) 0.16, 0.24, and 0.64 mL SC injection CAM2038 (buprenorphine FluidCrystal® once-weekly injection depot)
  CAM2038 q4w ( buprenorphine FluidCrystal®): SC injection depot for once monthly administration (356 mg/mL) at doses of 64, 96, 128 mg (buprenorphine base) 0.18, 0.27, and 0.36 mL SC injection CAM2038 (buprenorphine FluidCrystal® once-monthly injection depot)
- Placebo Subcutaneous Injections: CAM2038 placebo: 0.16, 0.18, 0.24, 0.27, 0.36, and 0.64 mL SC injection administered once weekly or once monthly (matching volumes for CAM2038 q1w and near-matching volumes for CAM2038 q4w).
Arm/Group | CAM2038 (Buprenorphine FluidCrystal®) q1w and q4w | Placebo Subcutaneous Injections
Number analyzed (Participants) | 112 | 110
score on a scale
  Baseline | 2.7 (1.26) | 2.4 (1.25)
  Change from Baseline to Week 12: number analyzed (Participants) | 75 | 69
  Change from Baseline to Week 12 | -0.9 (1.62) | -1.9 (1.97)

2. Primary Outcome: Change From Baseline in Weekly Average of (Daily) Average Pain Intensity (WAAPI) of the Open Label Phase.
Description: Change from baseline in Weekly Average of (Daily) Average Pain Intensity (WAAPI) of the Open Label Phase based on the 11-Point numerical rating scale with 10 being the worst pain. Baseline is defined as the last week prior to Visit 14 (Randomization Visit) for the roll-over subjects and the last week prior to Visit 14 (Enrollment Visit) for de novo subjects.
Time Frame: 48 weeks -From baseline to 48 weeks after baseline (Baseline is defined as the last week prior to Visit 14 (Randomization Visit) for the roll-over subjects and the last week prior to Visit 14 (Enrollment Visit) for de novo subjects).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- De Novo: CAM2038 50 mg/mL q1w at doses of 4 mg, 8 mg, 12 mg CAM2038 356 mg/mL q4w at doses of 64 mg, 96 mg, or 128 mg.
  buprenorphine
- CAM2038: CAM2038 50 mg/mL q1w at doses of 4 mg, 8 mg, 12 mg CAM2038 356 mg/mL q4w at doses of 64 mg, 96 mg, or 128 mg buprenorphine during both Double Blind Phase and Open Label Phase
- Rollover Placebo Injections: Placebo injections during Double Blind Phase, CAM2038 50 mg/mL q1w at doses of 4 mg, 8 mg, 12 mg orCAM2038 356 mg/mL q4w at doses of 64 mg, 96 mg, or 128 mg buprenorphine during Open Label Phase
Arm/Group | De Novo | CAM2038 | Rollover Placebo Injections
Number analyzed (Participants) | 54 | 24 | 31
score on a scale
  Baseline: number analyzed (Participants) | 54 | 21 | 31
  Baseline | 2.839 (1.0753) | 2.256 (1.1642) | 1.944 (1.1288)
  Change from Baseline to Week 4: number analyzed (Participants) | 50 | 21 | 31
  Change from Baseline to Week 4 | -0.434 (0.94) | -0.531 (0.93) | -1.586 (1.80)
  Change from Baseline to Week 8: number analyzed (Participants) | 50 | 21 | 31
  Change from Baseline to Week 8 | -0.555 (1.28) | -0.729 (0.99) | -2.165 (2.20)
  Change from Baseline to Week 12: number analyzed (Participants) | 47 | 20 | 30
  Change from Baseline to Week 12 | -0.752 (1.35) | -0.767 (1.20) | -2.079 (2.01)
  Change from Baseline to Week 16: number analyzed (Participants) | 45 | 15 | 27
  Change from Baseline to Week 16 | -0.543 (1.19) | -0.312 (0.68) | -1.229 (1.42)
  Change from Baseline to Week 20: number analyzed (Participants) | 44 | 18 | 26
  Change from Baseline to Week 20 | -0.690 (1.47) | -0.566 (1.05) | -1.013 (1.63)
  Change from Baseline to Week 24: number analyzed (Participants) | 45 | 18 | 25
  Change from Baseline to Week 24 | -0.718 (1.46) | -0.872 (1.51) | -1.220 (1.41)
  Change from Baseline to Week 28: number analyzed (Participants) | 43 | 17 | 25
  Change from Baseline to Week 28 | -0.905 (1.56) | -0.338 (1.06) | -1.212 (1.46)
  Change from Baseline to Week 32: number analyzed (Participants) | 42 | 17 | 27
  Change from Baseline to Week 32 | -0.941 (1.64) | -0.275 (1.41) | -1.111 (1.27)
  Change from Baseline to Week 36: number analyzed (Participants) | 40 | 17 | 26
  Change from Baseline to Week 36 | -0.920 (1.48) | -0.623 (1.36) | -1.119 (1.42)
  Change from Baseline to Week 40: number analyzed (Participants) | 41 | 17 | 25
  Change from Baseline to Week 40 | -0.913 (1.37) | -0.519 (1.51) | -1.113 (1.49)
  Change from Baseline to Week 44: number analyzed (Participants) | 38 | 15 | 22
  Change from Baseline to Week 44 | -0.767 (1.32) | -0.560 (1.37) | -1.282 (1.57)
  Change from Baseline to Week 48: number analyzed (Participants) | 32 | 15 | 14
  Change from Baseline to Week 48 | -0.996 (1.39) | -0.619 (1.58) | -1.215 (1.57)

3. Secondary Outcome: Change From Baseline in the Weekly Average of (Daily) Worst Pain Intensity Scores at Week 12 of the Double-Blind Phase Based on 11-Point Numerical Rating Scale With 10 Being the Worst Pain.
Description: Change from baseline in Weekly Average of (Daily) Worst Pain Intensity (WAWPI) and the primary timepoint will be Week 12 of the Double-Blind Phase based on the 11-Point numerical rating scale with 0 being no pain and 10 being the worst pain.
Time Frame: 12 weeks- from randomization baseline to 12 weeks after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CAM2038: CAM2038 50 mg/mL q1w at doses of 8 mg, 12 mg, CAM2038 356 mg/mL q4w at doses of 64 mg, 96 mg, or 128 mg.
  buprenorphine
- Placebo: CAM2038 placebo: 0.16, 0.18, 0.24, 0.27, 0.36, and 0.64 mL SC injection administered once weekly or once monthly (matching volumes for CAM2038 q1w and near-matching volumes for CAM2038 q4w).
Arm/Group | CAM2038 | Placebo
Number analyzed (Participants) | 112 | 110
score on a scale
  Baseline: number analyzed (Participants) | 109 | 110
  Baseline | 3.8 (1.59) | 3.7 (1.65)
  Change from Baseline to Week 12: number analyzed (Participants) | 76 | 69
  Change from Baseline to Week 12 | -1.1 (1.81) | -2.2 (2.18)

4. Secondary Outcome: Number of Subjects With a 30% and 50% Reduction in WAAPI From Baseline to Week 12 of the Double-Blind Phase.
Description: Number of Responders With a 30% and 50% Reduction in WAAPI from the Open-Label Titration Period Baseline to Week 12 of the Double-Blind Treatment Period (mITT Population)
Time Frame: 12 weeks- from randomization baseline to 12 weeks after randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- CAM2038: CAM2038 50 mg/mL q1w at doses of 8 mg, 12 mg, 16 mg, 24 mg, or 32 mg. CAM2038 356 mg/mL q4w at doses of 64 mg, 96 mg, or 128 mg.
  buprenorphine
- Placebo: CAM2038 placebo injections
  Placebo
Arm/Group | CAM2038 | Placebo
Number analyzed (Participants) | 112 | 110
Participants
  >= 30% improvement | 60 | 47
  >= 50% improvement | 44 | 32

5. Secondary Outcome: Summary of Rescue Medication Usage- Double-Blind Phase.
Description: Rescue medication usage (number of days used) during the Double-Blind Phase.
Time Frame: 12 weeks- from randomization baseline to 12 weeks after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CAM2038 | Placebo
Number analyzed (Participants) | 112 | 110
Days
  Baseline: number analyzed (Participants) | 109 | 110
  Baseline | 3.4 (2.84) | 3.5 (2.91)
  Change from Baseline to Week 12: number analyzed (Participants) | 77 | 70
  Change from Baseline to Week 12 | -1.5 (2.58) | -2.1 (2.63)

6. Secondary Outcome: Change From Open Label Titration Baseline to Week 12 of the Double-Blind Phase in EuroQol Group 5-dimension 5-level Self-report Questionnaire Score.
Description: Change from Open Label Titration baseline to Week 12 of the Double-Blind Phase in EuroQol Group 5-dimension 5-level self-report questionnaire score. The EuroQoL Group 5-Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) descriptive system is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows subjects to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood, using a 5-level scale. These combinations of attributes were converted into a weighted health-state index score, according to the US population-based algorithm, with higher scores indicating better quality of life. The score ranges from 0-100 with 0 as the worst health and 100 as the best health.
Time Frame: 12 weeks- from randomization baseline to 12 weeks after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CAM2038: CAM2038 50 mg/mL q1w at doses of 8 mg, 12 mg CAM2038 356 mg/mL q4w at doses of 64 mg, 96 mg, or 128 mg.
  buprenorphine
Arm/Group | CAM2038 | Placebo
Number analyzed (Participants) | 112 | 110
units on a scale
  Titration Baseline: number analyzed (Participants) | 112 | 106
  Titration Baseline | 63.7 (20.55) | 61.3 (22.05)
  Change from Baseline to Week 12: number analyzed (Participants) | 108 | 110
  Change from Baseline to Week 12 | -9.4 (18.47) | -7.2 (23.04)

7. Secondary Outcome: Change From Baseline to Week 12 of the Double-Blind Phase in Work Productivity and Activity Impairment Score
Description: Change from baseline to Week 12 of the Double-Blind Phase in Work Productivity and Activity Impairment score. The Work Productivity and Activity Impairment (WPAI) is a self-administered instrument used to measure the effect of general health and symptom severity on work productivity and regular activities, and yields 4 types of scores (higher scores indicate greater impairment): Absenteeism (work time missed)，Presenteeism (impairment at work/reduced on-the-job effectiveness), Work Productivity Loss (overall work impairment/absenteeism plus presenteeism)，and Activity Impairment. Scores range from 0-100 for each of the four types with higher scores indicating greater impairment.
Time Frame: 23 weeks- from baseline to 12 weeks after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAM2038 | Placebo
Number analyzed (Participants) | 112 | 110
score on a scale
  Baseline-Activity Impairment | 58.8 (23.68) | 61.2 (22.74)
  Change from Baseline to Week 12 after randomization-Activity impairment: number analyzed (Participants) | 108 | 106
  Change from Baseline to Week 12 after randomization-Activity impairment | 18.1 (24.88) | 11.7 (26.28)
  Baseline-Absenteesim: number analyzed (Participants) | 33 | 35
  Baseline-Absenteesim | 5.1 (10.19) | 9.9 (22.50)
  Change from Baseline to Week 12 after randomization-Absenteesim: number analyzed (Participants) | 30 | 29
  Change from Baseline to Week 12 after randomization-Absenteesim | -0.8 (10.75) | -4.6 (22.88)
  Baseline-Presenteeism: number analyzed (Participants) | 35 | 36
  Baseline-Presenteeism | 38.9 (22.33) | 47.8 (25.20)
  Change from Baseline to Week 12 after randomization-Presenteeism: number analyzed (Participants) | 32 | 31
  Change from Baseline to Week 12 after randomization-Presenteeism | 5.0 (27.47) | 9.0 (27.37)
  Baseline-Work Productivity Loss: number analyzed (Participants) | 33 | 35
  Baseline-Work Productivity Loss | 41.3 (23.09) | 52.3 (26.77)
  Change from Baseline to Week 12 after randomization- Work Productivity Loss: number analyzed (Participants) | 30 | 29
  Change from Baseline to Week 12 after randomization- Work Productivity Loss | 5.4 (23.05) | 7.8 (26.40)

8. Secondary Outcome: Number of Subjects Discontinued Due to Loss of Efficacy
Description: Number of Subjects Discontinued due to loss of efficacy, defined as discontinuation of study drug for lack of efficacy.
Time Frame: 12 weeks- from randomization baseline to 12 weeks after randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CAM2038 | Placebo
Number analyzed (Participants) | 112 | 110
Participants | 7 | 21

9. Secondary Outcome: Change From Baseline to Week 12 of the Double-Blind Phase in Patient Global Impression of Improvement (PGI-I) Scale
Description: Change from baseline to Week 12 of the Double-Blind Phase in Patient global Impression of Improvement (PGI-I) Scale. PGI-I)Scale is a single question 7-point likert scale that required the subject to assess how much his/her pain had improved or worsened relative to the start of the study at the beginning of the intervention . Ratings were: 1, much worse; 2, worse; 3, a little worse; 4, no change; 5, a little better; 6, better; or 7, much better
Time Frame: 12 weeks- from baseline (randomization) to 12 weeks after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAM2038 | Placebo
Number analyzed (Participants) | 112 | 110
units on a scale
  Baseline: number analyzed (Participants) | 111 | 110
  Baseline | 6.0 (0.96) | 6.2 (0.74)
  Change from Baseline to Week 12: number analyzed (Participants) | 107 | 106
  Change from Baseline to Week 12 | 0.4 (1.48) | 1.5 (1.63)

10. Secondary Outcome: Change From Baseline in Weekly Average of (Daily) Worst Pain Intensity (WAWPI) of the Open Label Phase.
Description: Change from baseline in Weekly Average of (Daily) Worst Pain Intensity (WAWPI) and the primary timepoint will be Week 52 of the Open Label Phase based on the 11-Point numerical rating scale with 10 being the worst pain. Baseline is defined as the last week prior to Visit 14 (Randomization Visit) for the roll-over subjects and the last week prior to Visit 14 (Enrollment Visit) for de novo subjects.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | De Novo | CAM2038 | Rollover Placebo Injections
Number analyzed (Participants) | 54 | 21 | 31
score on a scale
  Baseline | 4.139 (1.55) | 3.717 (3.86) | 3.246 (3.29)
  Change from Baseline to Week 4: number analyzed (Participants) | 50 | 21 | 31
  Change from Baseline to Week 4 | -0.517 (1.34) | -0.859 (1.57) | -1.734 (1.97)
  Change from Baseline to Week 8: number analyzed (Participants) | 50 | 21 | 31
  Change from Baseline to Week 8 | -0.625 (1.48) | -1.066 (1.68) | -2.404 (2.47)
  Change from Baseline to Week 12: number analyzed (Participants) | 47 | 20 | 30
  Change from Baseline to Week 12 | -0.846 (1.53) | -1.157 (1.95) | -2.455 (2.26)
  Change from Baseline to Week 16: number analyzed (Participants) | 45 | 15 | 27
  Change from Baseline to Week 16 | -0.689 (1.51) | -0.487 (1.14) | -1.587 (2.03)
  Change from Baseline to Week 20: number analyzed (Participants) | 44 | 18 | 26
  Change from Baseline to Week 20 | -0.725 (1.59) | -0.592 (1.157) | -1.391 (2.18)
  Change from Baseline to Week 24: number analyzed (Participants) | 45 | 18 | 25
  Change from Baseline to Week 24 | -0.735 (1.67) | -0.902 (2.13) | -1.461 (1.97)
  Change from Baseline to Week 28: number analyzed (Participants) | 43 | 17 | 25
  Change from Baseline to Week 28 | -1.013 (1.55) | -0.518 (1.74) | -1.531 (2.13)
  Change from Baseline to Week 32: number analyzed (Participants) | 42 | 17 | 27
  Change from Baseline to Week 32 | -0.996 (1.90) | -0.322 (1.76) | -1.462 (2.06)
  Change from Baseline to Week 36: number analyzed (Participants) | 40 | 17 | 26
  Change from Baseline to Week 36 | -1.044 (1.71) | -0.682 (0.20) | -1.112 (1.34)
  Change from Baseline to Week 40: number analyzed (Participants) | 41 | 17 | 25
  Change from Baseline to Week 40 | -0.935 (1.50) | -0.658 (1.92) | -1.087 (1.48)
  Change from Baseline to Week 44: number analyzed (Participants) | 38 | 15 | 22
  Change from Baseline to Week 44 | -0.897 (1.56) | -0.764 (2.03) | -1.216 (1.68)
  Change from Baseline to Week 48: number analyzed (Participants) | 32 | 15 | 18
  Change from Baseline to Week 48 | -1.059 (1.59) | -0.896 (2.26) | -1.292 (1.78)

11. Secondary Outcome: Subject Discontinued Due to Loss of Efficacy, Defined as Discontinuation of Study Drug for Lack of Efficacy.
Description: Subject Discontinued Due to Loss of Efficacy, Defined as Discontinuation of Study Drug for Lack of Efficacy Open Label Phase.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo | CAM2038 | Rollover Placebo Injections
Number analyzed (Participants) | 54 | 24 | 31
Participants | 1 | 0 | 1

12. Secondary Outcome: Summary of Rescue Medication Usage-Open Label Phase
Description: Rescue medication usage (number of days used) during the Open Label Phase.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | De Novo | CAM2038 | Rollover Placebo Injections
Number analyzed (Participants) | 54 | 24 | 31
Days
  Baseline: number analyzed (Participants) | 54 | 21 | 31
  Baseline | 1.172 (1.99) | 0.352 (0.68) | 1.330 (2.23)
  Change from Baseline to Week 4: number analyzed (Participants) | 50 | 21 | 31
  Change from Baseline to Week 4 | -0.744 (1.54) | -0.793 (2.47) | -1.124 (2.32)
  Change from Baseline to Week 8: number analyzed (Participants) | 50 | 21 | 31
  Change from Baseline to Week 8 | -0.301 (1.75) | -0.671 (2.18) | -1.672 (2.29)
  Change from Baseline to Week 12: number analyzed (Participants) | 47 | 20 | 30
  Change from Baseline to Week 12 | -0.472 (1.99) | -1.180 (2.48) | -1.817 (2.53)
  Change from Baseline to Week 16: number analyzed (Participants) | 45 | 15 | 27
  Change from Baseline to Week 16 | -0.679 (1.87) | -0.418 (2.33) | -0.990 (2.07)
  Change from Baseline to Week 20: number analyzed (Participants) | 44 | 18 | 26
  Change from Baseline to Week 20 | -0.562 (2.00) | -0.745 (2.02) | -0.490 (2.48)
  Change from Baseline to Week 24: number analyzed (Participants) | 45 | 18 | 25
  Change from Baseline to Week 24 | -0.689 (1.96) | -0.959 (2.52) | -0.933 (2.64)
  Change from Baseline to Week 28: number analyzed (Participants) | 43 | 17 | 25
  Change from Baseline to Week 28 | -1.045 (2.17) | -0.553 (1.64) | -0.875 (2.80)
  Change from Baseline to Week 32: number analyzed (Participants) | 42 | 17 | 27
  Change from Baseline to Week 32 | -0.864 (2.36) | -0.577 (2.12) | -1.280 (2.70)
  Change from Baseline to Week 36: number analyzed (Participants) | 40 | 17 | 26
  Change from Baseline to Week 36 | -0.989 (2.29) | -0.359 (1.63) | -1.479 (2.91)
  Change from Baseline to Week 40: number analyzed (Participants) | 41 | 17 | 25
  Change from Baseline to Week 40 | -0.941 (2.41) | -0.980 (2.26) | -1.339 (2.81)
  Change from Baseline to Week 44: number analyzed (Participants) | 38 | 15 | 22
  Change from Baseline to Week 44 | -1.050 (2.54) | -0.767 (1.90) | -1.465 (2.51)
  Change from Baseline to Week 48: number analyzed (Participants) | 32 | 15 | 18
  Change from Baseline to Week 48 | -1.088 (2.20) | -0.929 (2.15) | -2.302 (2.89)

13. Secondary Outcome: Summary of Change From Baseline in EuroQoL Group EQ-5D-5L Scores Over Time-Open Label Phase
Description: Change from Open Label Titration baseline in EuroQol Group 5-dimension 5-level self-report questionnaire score in the Open Label Phase. The EuroQoL Group 5-Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) descriptive system is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows subjects to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood, using a 5-level scale. These combinations of attributes were converted into a weighted health-state index score, according to the US population-based algorithm, with higher scores indicating better quality of life. The score ranges from 0-100 with 0 as the worst health and 100 as the best health.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | De Novo | CAM2038 | Rollover Placebo Injections
Number analyzed (Participants) | 54 | 24 | 31
score on a scale
  Baseline | 76.59 (13.31) | 83.38 (14.89) | 79.65 (14.00)
  Change from Baseline at End of Treatment Visit: number analyzed (Participants) | 52 | 24 | 31
  Change from Baseline at End of Treatment Visit | 5.17 (15.43) | 9.95 (18.83) | 6.35 (18.95)

14. Secondary Outcome: Summary of Change From Baseline in Clinical Global Impression of Improvement (CGI-I) Scale-Open Label
Description: Summary of Change from Baseline in Clinical Global Impression of Improvement (CGI-I) scale. The Clinician Global Impression of Improvement (CGI-I) Scale is a 7-point scale that required the clinician to assess how much the subject's Pain had improved or worsened relative to the start of the study. Assessments were rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | De Novo | CAM2038 | Rollover Placebo Injections
Number analyzed (Participants) | 54 | 24 | 31
score on a scale
  Baseline: number analyzed (Participants) | 53 | 24 | 30
  Baseline | 1.9 (0.79) | 1.7 (0.56) | 2.0 (1.13)
  Change from Baseline at End of Treatment Visit | -0.4 (1.25) | -0.1 (1.08) | 0.1 (1.31)

15. Secondary Outcome: Summary of Change From Baseline in Patient Global Impression of Improvement (PGI-I) Scale
Description: Change from baseline in the Open Label Phase in Patient global Impression of Improvement (PGI-I) Scale. PGI-I Scale is a single question 7-point likert scale that required the subject to assess how much his/her pain had improved or worsened relative to the start of the study. Ratings were: 1, much worse; 2, worse; 3, a little worse; 4, no change; 5, a little better; 6, better; or 7, much better
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | De Novo | CAM2038 | Rollover Placebo Injections
Number analyzed (Participants) | 54 | 24 | 31
score on a scale
  Baseline: number analyzed (Participants) | 38 | 20 | 28
  Baseline | 5.8 (0.84) | 6.1 (1.10) | 6.3 (0.84)
  Change from Baseline at End of Treatment Visit | 0.2 (1.16) | -0.2 (1.04) | 0.5 (0.92)

16. Secondary Outcome: Summary of Change From Baseline in Work Productivity and Activity Impairment Questionnaire (WPAI) Open Label Phase
Description: Change from baseline in the Open Label Phase in Work Productivity and Activity Impairment score with a range of 0-100 for 4 types of scores with higher scores indicating greater impairment. The Work Productivity and Activity Impairment (WPAI) is a self-administered instrument used to measure the effect of general health and symptom severity on work productivity and regular activities, and yields 4 types of scores (higher scores indicate greater impairment): Absenteeism (work time missed)，Presenteeism (impairment at work/reduced on-the-job effectiveness), Work Productivity Loss (overall work impairment/absenteeism plus presenteeism)，and Activity Impairment. Scores range from 0-100 for each of the four types with higher scores indicating greater impairment.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | De Novo | CAM2038 | Rollover Placebo Injections
Number analyzed (Participants) | 54 | 24 | 31
score on a scale
  Baseline-Absenteesim: number analyzed (Participants) | 13 | 7 | 10
  Baseline-Absenteesim | 1.538 (5.55) | 0 (0) | 0 (0)
  Change from Baseline at End of Treatment Visit-Absenteesim: number analyzed (Participants) | 10 | 6 | 9
  Change from Baseline at End of Treatment Visit-Absenteesim | 0 (0) | -2.137 (5.23) | 0 (0)
  Baseline-Presenteeism: number analyzed (Participants) | 13 | 7 | 10
  Baseline-Presenteeism | 26.9 (18.43) | 22.9 (19.76) | 21.0 (11.97)
  Change from Baseline at End of Treatment Visit-Presenteeism | 1.0 (15.95) | 1.7 (7.53) | 6.7 (23.98)
  Baseline-Work Productivity Loss: number analyzed (Participants) | 13 | 7 | 10
  Baseline-Work Productivity Loss | 27.846 (19.42) | 22.857 (19.76) | 21.000 (11.97)
  Change from Baseline at End of Treatment Visit- Work Productivity Loss: number analyzed (Participants) | 10 | 6 | 9
  Change from Baseline at End of Treatment Visit- Work Productivity Loss | 1.000 (15.95) | -0.043 (11.05) | 6.667 (23.98)
  Baseline-Activity Impairment: number analyzed (Participants) | 38 | 20 | 28
  Baseline-Activity Impairment | 32.1 (20.55) | 29.0 (23.82) | 22.9 (16.52)
  Change from Baseline at End of Treatment Visit-Activity Impairment: number analyzed (Participants) | 38 | 20 | 28
  Change from Baseline at End of Treatment Visit-Activity Impairment | -12.1 (22.20) | -6.5 (25.60) | -18.2 (22.45)

17. Secondary Outcome: Number of Subjects Discontinued Due to Loss of Efficacy
Description: Number of Subjects Discontinued due to loss of efficacy, defined as discontinuation of study drug for lack of efficacy.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo | CAM2038 | Rollover Placebo Injections
Number analyzed (Participants) | 54 | 24 | 31
Participants | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Double Blind Phase-up to 26 weeks Open Label Phase-up to 64 weeks
Groups:
- CAM2038 q1w or q4w BPN Treatment-Titration Period of Double Blind Phase; De Novo Subjects-Open Label, Titration Period Only: CAM2038 q1w (buprenorphine FluidCrystal®) : SC injection depot for once weekly or monthly administration at doses of 4, 8, 12, 16, 24 and 32 mg (buprenorphine base) 0.16, 0.24, and 0.64 mL SC injection CAM2038 (buprenorphine FluidCrystal® once-weekly injection depot)
- CAM2038 q1w or q4w BPN Treatment- Double Blind Period of Double Blind Phase: CAM2038 50 mg/mL q1w at doses of 4, mg 8 mg, 12 mg, CAM2038 356 mg/mL q4w at doses of 64 mg, 96 mg, or 128 mg. buprenorphine
- Placebo Subcutaneous Injections-Double Blind Period of Double Blind Phase: CAM2038 placebo: 0.16, 0.18, 0.24, 0.27, 0.36, and 0.64 mL SC injection administered once weekly or once monthly (matching volumes for CAM2038 q1w and near-matching volumes for CAM2038 q4w).
- Rollover Subjects-Open Label, Titration Period Only: CAM2038 q1w (buprenorphine FluidCrystal®) : SC injection depot for once weekly or monthly administration at doses of 4, 8, 12, 16, 24 and 32 mg (buprenorphine base) 0.16, 0.24, and 0.64 mL SC injection
- De Novo Subjects-Open Label, Enrollment Period Only; Rollover Subjects-Open Label, Enrollment Period Only: CAM2038 q1w (buprenorphine FluidCrystal®) : SC injection depot for once weekly or monthly administration at doses of 4, 8, 12 mg (buprenorphine base) 0.16, 0.24, and 0.64 mL SC injection CAM2038 (buprenorphine FluidCrystal® once-weekly injection depot)
  CAM2038 q4w ( buprenorphine FluidCrystal®): SC injection depot for once monthly administration (356 mg/mL) at doses of 64, 96, 128 mg (buprenorphine base) 0.18, 0.27, and 0.36 mL SC injection CAM2038 (buprenorphine FluidCrystal® once-monthly injection depot)
Arm/Group | CAM2038 q1w or q4w BPN Treatment-Titration Period of Double Blind Phase | CAM2038 q1w or q4w BPN Treatment- Double Blind Period of Double Blind Phase | Placebo Subcutaneous Injections-Double Blind Period of Double Blind Phase | De Novo Subjects-Open Label, Titration Period Only | Rollover Subjects-Open Label, Titration Period Only | De Novo Subjects-Open Label, Enrollment Period Only | Rollover Subjects-Open Label, Enrollment Period Only
All-Cause Mortality (participants affected / at risk) | 1/468 | 0/112 | 1/110 | 0/75 | 0/46 | 0/54 | 0/55
Serious Adverse Events (participants affected / at risk) | 10/468 | 3/112 | 3/110 | 1/75 | 1/46 | 7/54 | 7/55
Other Adverse Events (participants affected / at risk) | 300/468 | 36/112 | 32/110 | 41/75 | 15/46 | 41/54 | 46/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAM2038 q1w or q4w BPN Treatment-Titration Period of Double Blind Phase (N=468) | CAM2038 q1w or q4w BPN Treatment- Double Blind Period of Double Blind Phase (N=112) | Placebo Subcutaneous Injections-Double Blind Period of Double Blind Phase (N=110) | De Novo Subjects-Open Label, Titration Period Only (N=75) | Rollover Subjects-Open Label, Titration Period Only (N=46) | De Novo Subjects-Open Label, Enrollment Period Only (N=54) | Rollover Subjects-Open Label, Enrollment Period Only (N=55)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizzyness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAM2038 q1w or q4w BPN Treatment-Titration Period of Double Blind Phase (N=468) | CAM2038 q1w or q4w BPN Treatment- Double Blind Period of Double Blind Phase (N=112) | Placebo Subcutaneous Injections-Double Blind Period of Double Blind Phase (N=110) | De Novo Subjects-Open Label, Titration Period Only (N=75) | Rollover Subjects-Open Label, Titration Period Only (N=46) | De Novo Subjects-Open Label, Enrollment Period Only (N=54) | Rollover Subjects-Open Label, Enrollment Period Only (N=55)
Constipation (Gastrointestinal disorders) | 25 (25) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 87 (87) | 2 (2) | 1 (1) | 9 (9) | 7 (7) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 64 (64) | 3 (3) | 1 (1) | 7 (7) | 4 (4) | 3 (3) | 3 (3)
Injection Site Erythema (General disorders) | 32 (32) | 2 (2) | 3 (3) | 6 (6) | 0 (0) | 1 (1) | 3 (3)
Injection site pain (General disorders) | 29 (29) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 2 (2) | 1 (1)
Injection site pruritus (General disorders) | 40 (40) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 2 (2) | 3 (3)
Injection Site Swelling (General disorders) | 25 (25) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
Upper respiratory tract injection (Infections and infestations) | 6 (6) | 2 (2) | 4 (4) | 6 (6) | 1 (1) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Nasopharyngitis (Infections and infestations) | 7 (7) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 8 (8) | 5 (5) | 7 (7) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 16 (16) | 5 (5) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (15) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 6 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 7 (7) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 38 (38) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 28 (28) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT02946073/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT02946073/SAP_001.pdf